CLINICAL TRIAL: NCT01778205
Title: Phase 1 Study of the Effect of Maternal Nutritional Status on Placental Vascular Function, Fetal Growth and Intrauterine Growth Retardation.
Brief Title: The Reus-Tarragona Birth Cohort Study of Early Development and Ageing.
Status: Completed | Type: Observational
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Italfarmaco (Industry); Instituto de Salud Carlos III (Other Government); State Research Agency, Spain (Other Government); JPI ERA-HDHL (Unknown); University Rovira i Virgili (Other); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Dr. Michelle Murphy, Profesora agregat, Institut Investigacio Sanitaria Pere Virgili
Other Study IDs: IISPV_Murphy1; SPAIN MICINN (Other Grant/Funding Number: Ministerio de Ciéncia y Innovación SAF2005/05096); SPAIN ISCIII (Other Grant/Funding Number: Instituto de Salud Carlos III PI10/00335); SPAIN URV (Other Grant/Funding Number: Universitat Rovira i Virgili); SPAIN ISCIII (Other Grant/Funding Number: Instituto de Salud Carlos III PI13/02500); SPAIN ISCIII (Other Grant/Funding Number: Instituto de Salud Carlos III PI19/00844); SPAIN AEI (Other Grant/Funding Number: Agencia Estatal Investigacion PCI2018-093098); Horizon 2020 (Other Grant/Funding Number: JPI ERA-HDHL Nutrition & The Epigenome)
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Intrauterine Development
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Serum Leukocytes Placenta
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women with confirmed viable fetus at first prenatal check-up at <12 gestational weeks
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational

SUMMARY:
The recent fall in birth and death rates has led to demographic changes such as low fertility and high life expectancy . The WHO reports the median age of the European population to be the highest in the world and predicts that the proportion of over-60s in will increase from 14% in 2010 to 25% in 2050. There is wide variability in the quality of health and well-being in the ageing population. Longevity with a good quality of life is a consequence of the combination of an individual's genes, nutrition, environment, lifestyle and medical interventions. There is increasing evidence that research into healthy ageing needs to start with early life data to capture all traits and exposures experienced by an individual throughout life. Epigenetic imprinting occurs both in utero and during early postnatal development. Maternal environmental exposures, including nutritional status, may have a permanent effect on the developing foetus by influencing epigenetic profiles and leading to life-long genome adaptation. Numerous reports show that restricted intra-uterine growth due to poor maternal nutrition during pregnancy increases risk in the offspring of developing mental disorders, metabolic syndrome, cardiovascular disease or stroke in later life. To understand the basic mechanisms and interactions through which the ageing phenotype develops, systems involved in key processes of early development must be considered as well as those crucial to health in older persons. The Reus and Tarragona Birth Cohort is a longitudinal study. In the first phase, blood is collected from pregnant women at <12, 15, 24-27 and 34 gestational weeks (GW) and at labor and from the cord. Detailed lifestyle, habits and supplement use data are collected at 20 and 32 gestational weeks and on nutritional habits at <12GW and at birth. Placental vascular function is assessed at 20 and 32 GW by analysis of Doppler waveforms of the uterine arteries. Data on pregnancy evolution and outcome are also recorded. The first phase investigates the association between gene-environment (nutrient and lifestyle habits) interactions and fetal growth and pregnancy outcome. The second phase of the study follows up the children at 7.5 years of age. Growth, exercise and nutritional habits as well as environment and cognitive development are assessed. The aims are to investigate the association between gene-environment interactions associated with healthy development from early pregnancy until 7.5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* <12 weeks pregnant at first prenatal check up

Exclusion Criteria:

* Illnesses / interventions affecting nutritional status, major recent surgery in the previous 6 months, multiple pregnancies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women less than 12 weeks pregnant at their first pre-natal check up are recruited from the URV University Hospitals: Sant Joan (Reus) and Joan XXIII (Tarragona)
Sampling Method: Non-Probability Sample
Enrollment: 831 (Actual)
Dates: Start 2005-01; Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Birth weight | At birth
Doppler waveforms of uterine arteries | 20 gestational weeks

OTHER OUTCOMES:
1-C metabolites | <12, 15, 24-27, 34 gestational weeks, at labor, in the cord
Intrauterine growth retardation | At birth

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Murphy, PhD, Principal Investigator — University Rovira i Virgili; Pere Cavallé-Busquets, MD, PHD, Study Director — Hospital Universitari Sant Joan de Reus; Joan D Fernandez-Ballart, PhD, Study Chair — University Rovira i Virgili; Mónica Ballesteros, MD, PHD, Study Director — Hospital de Tarragona Joan XXIII
Locations (2):
- Spain (2):
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital de Tarragona Joan XXIII, Tarragona

REFERENCES:
- [Background] Colomina JM, Cavalle-Busquets P, Fernandez-Roig S, Sole-Navais P, Fernandez-Ballart JD, Ballesteros M, Ueland PM, Meyer K, Murphy MM. Maternal Folate Status and the BHMT c.716G>A Polymorphism Affect the Betaine Dimethylglycine Pathway during Pregnancy. Nutrients. 2016 Oct 9;8(10):621. doi: 10.3390/nu8100621. PMID 27735840
- [Background] Sole-Navais P, Salat-Batlle J, Cavalle-Busquets P, Fernandez-Ballart J, Ueland PM, Ballesteros M, Ornosa-Martin G, Ingles-Puig M, Colomina JM, Murphy MM. Early pregnancy folate-cobalamin interactions and their effects on cobalamin status and hematologic variables throughout pregnancy. Am J Clin Nutr. 2018 Feb 1;107(2):173-182. doi: 10.1093/ajcn/nqx041. PMID 29529156
- [Background] Roige-Castellvi J, Murphy M, Hernandez-Martinez C, Sole-Navais P, Cavalle-Busquets P, Fernandez-Ballart J, Ballesteros M, Canals J. The effect of prenatal smoke exposure on child neuropsychological function: a prospective mother-child cohort study. J Reprod Infant Psychol. 2020 Feb;38(1):25-37. doi: 10.1080/02646838.2019.1580350. Epub 2019 Feb 19. PMID 30777448
- [Background] Cavalle-Busquets P, Ingles-Puig M, Fernandez-Ballart JD, Haro-Barcelo J, Rojas-Gomez A, Ramos-Rodriguez C, Ballesteros M, Meyer K, Ueland PM, Murphy MM. Moderately elevated first trimester fasting plasma total homocysteine is associated with increased probability of miscarriage. The Reus-Tarragona Birth Cohort Study. Biochimie. 2020 Jun;173:62-67. doi: 10.1016/j.biochi.2020.01.008. Epub 2020 Jan 18. PMID 31962182
- [Result] Fernandez-Roig S, Cavalle-Busquets P, Fernandez-Ballart JD, Ballesteros M, Berrocal-Zaragoza MI, Salat-Batlle J, Ueland PM, Murphy MM. Low folate status enhances pregnancy changes in plasma betaine and dimethylglycine concentrations and the association between betaine and homocysteine. Am J Clin Nutr. 2013 Jun;97(6):1252-9. doi: 10.3945/ajcn.112.054189. Epub 2013 Apr 17. PMID 23595875
- [Derived] Santos-Calderon LA, Cavalle-Busquets P, Ramos-Rodriguez C, Grifoll C, Rojas-Gomez A, Ballesteros M, Ueland PM, Murphy MM. Folate and cobalamin status, indicators, modulators, interactions, and reference ranges from early pregnancy until birth: the Reus-Tarragona birth cohort study. Am J Clin Nutr. 2024 Nov;120(5):1269-1283. doi: 10.1016/j.ajcnut.2024.09.015. Epub 2024 Sep 24. PMID 39326699